CLINICAL TRIAL: NCT06959979
Title: Novel Molecular Targets and Innovative Therapeutic Perspective in Medulloblastoma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: University of Rome Tor Vergata (Other); Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello (Other); Università degli Studi di Enna Kore (Unknown)
Responsible Party: Principal Investigator, Tamburrini Gianpiero, Prof., Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PNRR-TR1-2023-12378243
Record Dates: First submitted 2024-07-24; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2024-07

CONDITIONS: Medulloblastoma, Childhood
MeSH Terms: conditions — Medulloblastoma | interventions — palbociclib; ribociclib; abemaciclib

STUDY DESIGN:
Intervention Model Description: Prospective, non-drug, non-device interventional study with molecular analysis on biological samples including a retrospective component. No patient procedures will be performed other than those within standard clinical practice. Specifically, the tumor will be collected during surgical removal and partially processed for organoid development, with the remainder stored for subsequent molecular comparisons between the organoid and the original tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prospective (Experimental): To establish ex-vivo translational models of MB, we will develop patient-derived organoids (PDOs) from primary surgical biopsies of patients
  Interventions: Drug: CDK4/6 Inhibitor (Palbociclib, Ribociclib, Abemaciclib)
- Retrospective (Experimental): To establish ex-vivo translational models of MB, we will develop patient-derived organoids (PDOs) from primary surgical biopsies of patients
  Interventions: Drug: CDK4/6 Inhibitor (Palbociclib, Ribociclib, Abemaciclib)

INTERVENTIONS:
Drug: CDK4/6 Inhibitor (Palbociclib, Ribociclib, Abemaciclib) — Evaluation of the response to CDK4/6 inhibitors (Palbociclib, Ribociclib, Abemaciclib) on selected Medulloblastoma (MB) patient-derived organoids (PDOs).
  Other Names: We will then evaluate the effects of CDK4/6 inhibitors on the selected MB PDOs.

SUMMARY:
Medulloblastoma (MB), a rare yet critical pediatric brain tumor, is divided into 4 molecular subgroups (WNT, SHH, Group 3, Group 4), each with distinct genetic profiles. Despite diagnostic and therapeutic advances, neurotoxicity from standard treatments (resection, radiotherapy, chemotherapy) and the need for long-term care remain challenges. CDK4/6 inhibitors (palbociclib, ribociclib, abemaciclib), approved for breast cancer, show potential in other tumors, but their efficacy in MB is unclear. Treatment resistance is a concern. This project aims to identify genetic markers of sensitivity to CDK4/6 inhibitors in MB, to improve therapies and overcome resistance.

DETAILED DESCRIPTION:
In this project, combining high-throughput molecular biology and translational approaches, we aim to identify the genetic and transcriptomic signatures that influence primary sensitivity and acquired resistance to CDK4/6 inhibitors in MB. Several key genetic events have been identified as determinants in MB. For example, MYC is among the most frequently amplified and best characterized oncogenes in G3-MB, a highly aggressive form of MB. PTCH1 or SUFU (negative regulators of the SHH signaling pathway) are recurrently mutated in SHH-MB, both in the germline and somatically, supporting a causal role for SHH signaling in these tumors. On the other hand, somatic mutations in CTNNB1 have been observed in patients with WNT-MB, leading to the activation of the WNT signaling pathway. Mutations in the CDK4/6 pathway also play an important role in the development of MB and are associated with poor outcomes for patients. It is important to emphasize that both the MYC pathway and the cyclin CDK4/6 RB pathway, which are frequently altered in MB, control the key cell fate decision to replicate the genome. For this reason, cell cycle regulators, such as CDK4/6 inhibitors, are currently considered attractive therapeutic targets. We have previously shown that the E3-ligase substrate receptor and autophagy regulator AMBRA1 promotes unrestricted CDK4/6 activity and confers resistance to palbociclib treatment in a wide range of tumors. Furthermore, our preliminary results suggest that the genetic alterations that drive MB onset influence the efficacy of CDK4/6 inhibitors. In this project, we aim to identify the genes and biological processes involved in the response to CDK4/6 inhibitors and to determine their relevance to MB.

Specific Aim 1: Genome-wide CRISPR/cas9 knockout screening of sensitivity to CDK4/6 inhibitors in MB. Recent studies have shown that cell cycle disruption is a key factor in MB onset and relapse. However, a unifying molecular mechanism involved in this process is still lacking. Furthermore, many of the therapeutic approaches that are under study in clinical trials lack solid molecular bases for systematic patient stratification. To fill this knowledge gap, we propose to develop an unbiased approach to identify genes that influence sensitivity to CDK4/6 inhibitors (palbociclib and abemaciclib). This approach will also help us better understand the regulatory networks that control progression and aggressiveness. We will use CRISPR/Cas9 technology to perform a genome-wide knockout (KO) screen. To this end, we will use the Human GeCKO v2 Pooled Knockout CRISPR library in MB cell lines expressing Cas9 ONS76 (SHH-MB), D283-MED (G3-MB) and HD-MB03 (G3-MB). These cell lines are representative of two distinct MB subgroups and also share p53 competence. This feature is relevant in the context of CDK4/6 inhibitors, because their efficacy strictly depends on the ability of p53 to induce senescence and cell cycle arrest. Cells will be treated or not with palbociclib and abemaciclib and maintained in log-growth phase at a 1000x coverage for sgRNA throughout the screen. The doses of palbociclib (0.07 μM) and abemaciclib (0.19 μM) were chosen as those that cause a 50% reduction in proliferation rate by cell count assays. After 14 days of treatment, genomic DNA will be extracted from each population and sgRNA sequencing libraries will be prepared. Identified genes will be ranked based on the protective effect that their KO exerts in both treated conditions. Subsequently, we will further characterize the top 5 non-redundant genes of interest (GOIs) that confer a growth advantage by biochemical and molecular biology approaches. In detail, we will assess the ability of GOIs to modulate the cell cycle by quantitative image-based cytometry (QIBC) and flow cytometry, in basal condition or upon CDK4/6 inhibition. To extend our results, we will validate the selected GOIs in other MB cell lines that we routinely use for cell biology assays (DAOY, D341-MED, CHLA-MED-01). Furthermore, we will implement our analysis by exploiting two cell lines (DAOY and ONS76) that we have already engineered to express two fluorescent reporters: FUCCI CA and DHB mVenere-p2a-mCherry-CDK4KTR. The former is a sophisticated technology that discriminates between cell cycle phases in a spatio-temporal manner using a double color combination. The latter is a reporter system that allows simultaneous monitoring of CDK4/6 and CDK2 activities in single cells. GOIs will be deleted in these cell lines by CRISPR/Cas9 technology and the effect of their ablation on cell growth and CDK4/6 inhibition will be studied. To gain mechanistic insights into how GOIs confer resistance to CDK4/6 inhibitors and to evaluate whether they enable acquired resistance, we will use an orthogonal approach to the CRISPR/Cas9 screen. We will develop in vitro models of acquired resistance by treating our panel of MB cells with abemaciclib or palbociclib. We will then perform RNA-seq to investigate whether the GOIs, or the pathways to which they belong, are modulated in resistant cells. Furthermore, since altering pre-mRNA processing regulation by treatment with an arginine methyltransferase PRMT5 inhibitor (GSK3326595) has recently been shown to restore sensitivity to palbociclib in tumor cells that have acquired resistance to this drug, we will test the combination of CDK4/6 inhibitors and PRMT5 in resistant MB cells.

Specific Aim 2: To establish ex-vivo translational models of MB, we will develop patient-derived organoids (PDOs) from primary surgical biopsies of patients. To this end, the Organoid Research Core Facility available at the P.I.'s Research Entity will be instrumental. Surgical biopsies will be enzymatically and mechanically digested and the tumor cell suspension (1x106 cells) will be mixed with Matrigel, allowed to assemble for 15 minutes at 37 °C and then seeded in tissue culture plates. Tumor organoids will be allowed to form for 4 days in culture in a humidified incubator at 37 °C. At the end of this incubation, tumor organoids will be transferred to an orbital shaker and will be cultured under agitation conditions (70 rpm) until passage for experimental assays. Once established, SHH-MB and G3-MB PDOs will be tested for their ability to capture the oncogenic characteristics of the original tumor. First, we will perform parallel immunohistochemical characterization of MB markers currently used for subtype specification in clinical practice. Subsequently, MB PDOs and original tissues will be sequenced to determine the mutational status of >500 genes frequently altered in human tumors using the TSO-500 (Illumina), as recently published at our Organoids Facility. Only PDOs that recapitulate the histological and genetic characteristics of the original tumor will be further propagated and used for functional studies. We will then evaluate the effects of CDK4/6 inhibitors on selected MB PDOs. Since these cell models grow in 3D and not all cells are directly accessible to the compounds delivered in the medium, we will first assess the cellular uptake and localization of palbociclib and abemaciclib. Since these compounds can be accumulated in lysosomes and other acidic cellular compartments, we will analyze the cellular uptake of CDK4/6 inhibitors in PDOs using the fluorescent properties of these drugs (~500 nm when excited at 405 nm light) in combination with fluorescent dyes used to label organelles in vivo (e.g., lysotracker, mitotracker). Subsequently, the impact of drug localization will be assessed by determining the proliferation, survival and senescence of PDOs in response to selected doses of CDK4/6 inhibitors using methods already in use at our facility. Furthermore, since the establishment and maintenance of PDOs depend on the presence of stem cells and stemness contributes to chemoresistance in MB, we will evaluate the effects of treatments on PDO stemness/differentiation characteristics by PCR and western blot analysis of previously established markers (CD133, Nestin, SOX1/2 for stemness; GFAP, CD44 for astrocytes; CD24, ßIII-tubulin for neuronal progenitors and neurons, respectively). PDOs sensitive to these drugs will then be cultured with suboptimal doses of CDK4/6 inhibitors for 2 months in order to select clones that acquire resistance to the treatments. RNA sequencing analyses of parental and CDK4/6-resistant PDOs will be performed and compared with the results obtained with MB cell lines (Specific Aim 1). Resistant PDOs will then be treated with CDK4/6 inhibitors with or without the PRMT5 inhibitor. Furthermore, the GOIs selected in Specific Aim 1 will be silenced in resistant PDOs by electroporation of sequence-specific siRNAs or CRISPR/Cas9 sgRNAs and the effects on sensitivity to CDK4/6 inhibitors will be evaluated. These studies will validate the functional relevance of GOIs and PRMT5 inhibition in a clinically relevant disease model.

Specific Aim 3: Development of innovative technologies for the evaluation of new clinical biomarkers for diagnosis and prognosis. To investigate the correlation between the GOIs selected in Specific Aims 1 and 2 and clinical parameters, we will analyze their expression in histological samples from MB patients. To this end, we will use the tissue slides from MB patients (n=60) that are stored at the UO1 Hospital and for which clinical follow-up is available. To date, immunohistochemistry (IHC) is the only clinically validated and commercially available approach to detect the distribution and amount of proteins in tissues by specific antigen-antibody reactions. However, IHC suffers from some drawbacks when new genes are under investigation. First, antibody production requires time-consuming processes that can lead to high analysis costs. Second, IHC involves several steps that affect the turnaround time of the technique. To overcome these limitations, we propose an alternative approach based on the use of synthetic DNA-based nanoswitches. More specifically, we will develop and characterize DNA nanoswitches capable of responding to specific proteins through a conformational change mechanism. Nanoswitches are composed of single-stranded DNA molecules (20-40 nucleotides) that serve as molecular scaffolds for the conjugation of different recognitions (protein epitopes, antibodies, aptamers) and signaling labels (fluorophore, quencher tag). The recognition will confer to the nanoswitch the ability to specifically bind to the protein of interest. The fluorophore/quencher pair will instead allow the signaling of the binding event. Nanoswitches are rationally designed to undergo a change upon binding to the protein of interest. This conformational change will force the fluorophore to move away from the quencher, leading to an increase in signal. This approach offers several advantages. Nanoswitches provide a signal only upon binding to the target protein, no washing and reaction steps are required. Nanoswitches are also versatile and can be labeled with different fluorophores, allowing for the orthogonal detection of several proteins simultaneously in the same sample.

In summary, this project aims to thoroughly investigate the role of CDK4/6 inhibitors in medulloblastoma (MB) treatment. By combining high-throughput molecular biology techniques with translational approaches, we will identify genetic and transcriptomic signatures that influence sensitivity and resistance to these inhibitors. We will also develop and utilize patient-derived organoids (PDOs) to validate our findings in a clinically relevant context. Furthermore, we will create innovative diagnostic tools using DNA nanoswitches to improve the detection of key biomarkers in MB. These studies have the potential to significantly advance our understanding of MB biology and pave the way for more effective and personalized treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* All patients affected by Medulloblastoma operated on at the Pediatric Neurosurgery Unit during their pediatric age will be elected to take part to the study

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Clarify the molecular mechanisms underlying the acquisition of resistance to CDK4/6i in MB. | 2 yrs
  Genetic characterization of PDOs derived from patients with medulloblastoma (MB).
  Measurement: Analysis of the mutational status of over 500 genes using TSO-500 sequencing, comparing the genetic profiles of PDOs with those of primary tumors.
Clarify the molecular mechanisms underlying the acquisition of resistance to CDK4/6i in MB. | 2 years
  Assessment of changes in cell proliferation in patient-derived organoids (PDOs) from medulloblastoma (MB) treated with CDK4/6 inhibitors compared to untreated controls.
  Measurement: Quantified by cell counting assays.
Clarify the molecular mechanisms underlying the acquisition of resistance to CDK4/6 inhibitors in medulloblastoma (MB). | 2 years
  Histological characterization of PDOs derived from patients with medulloblastoma (MB).
  Measurement: Evaluation of the expression of MB-specific histological markers by immunohistochemistry, comparing expression patterns between PDOs and primary tumors.
Clarify the molecular mechanisms underlying the acquisition of resistance to CDK4/6i in MB. | 2 years
  Assessment of changes in cell survival in patient-derived organoids (PDOs) from medulloblastoma (MB) treated with CDK4/6 inhibitors compared to untreated controls.
  Measurement: Quantified by cell viability assays.
Clarify the molecular mechanisms underlying the acquisition of resistance to CDK4/6i in MB. | 2 years
  Assessment of changes in cellular senescence levels in patient-derived organoids (PDOs) from medulloblastoma (MB) treated with CDK4/6 inhibitors compared to untreated controls.
  Measurement: Evaluated by analysis of senescence markers.
Clarify the molecular mechanisms underlying the acquisition of resistance to CDK4/6i in MB. | 2 years
  Outcome Measure Title: Quantitative change in cell proliferation Description: Quantitative change in cell proliferation expressed as a percentage variation from baseline.
  Unit of Measure: Percent change from baseline (%).
Clarify the molecular mechanisms underlying the acquisition of resistance to CDK4/6i in MB. | 2 years
  Outcome Measure Title: Quantitative change in cell survival Description: Quantitative change in cell survival expressed as a percentage variation from baseline.
  Unit of Measure: Percent change from baseline (%).
Clarify the molecular mechanisms underlying the acquisition of resistance to CDK4/6i in MB. | 2 years
  Outcome Measure Title: Quantitative change in cellular senescence Description: Quantitative change in cellular senescence expressed as a percentage variation from baseline.
  Unit of Measure: Percent change from baseline (%).

SECONDARY OUTCOMES:
CDK4/6 inhibitor-resistant clones | 2 years
  Proportion of medulloblastoma PDOs with maintained proliferation following exposure to CDK4/6 inhibitors, as assessed by cell viability assays.
transcriptomic analysis | 2 years
  Gene expression differences among medulloblastoma PDOs that are sensitive, primarily resistant, or secondarily resistant to CDK4/6 inhibitors.
Evaluate new therapeutic strategies | 2 years
  Reduction in cell viability of CDK4/6 inhibitor-resistant medulloblastoma PDOs following treatment with novel therapeutic combinations
Quantification of fluorescence intensity for tumor marker detection using synthetic DNA nanoswitches in histological sections from medulloblastoma patients and patient-derived organoids (PDOs) | 2 years
  Fluorescence intensity corresponding to specific tumor markers detected by synthetic DNA nanoswitches will be measured in histological sections of medulloblastoma patient tumors and patient-derived organoids (PDOs), using standardized fluorescence microscopy protocols.
  Measurement Tool: Fluorescence microscopy analysis (mean fluorescence intensity per sample).
  Unit of Measure: Mean fluorescence intensity (arbitrary fluorescence units, AFU).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Gemelli Irccs, Roma, ROMA, Italy

IPD SHARING:
Plan to Share IPD: No